CLINICAL TRIAL: NCT04942210
Title: Controlled Study of Immunogenicity and Safety of the Investigational vYF Candidate Vaccine in Comparison to YF-VAX in Adults
Brief Title: Study on an Investigational Yellow Fever Vaccine Compared With YF-VAX in Adults in the USA
Acronym: VYF02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYF02; U1111-1261-5612 (Registry Identifier: ICTRP); VYF02 (Other: Sanofi Identifier)
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Yellow Fever; Healthy Volunteers
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be performed in a modified double-blind fashion: Investigators, Sponsor, and study staff who conduct the safety assessment and the participant will not know which vaccine is administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- vYF (Experimental): 1 injection of vYF at Day 1
  Interventions: Biological: Yellow fever vaccine (produced on serum-free Vero cells)
- YF-VAX (Active Comparator): 1 injection of YF-VAX at Day 1
  Interventions: Biological: Yellow fever vaccine

INTERVENTIONS:
Biological: Yellow fever vaccine (produced on serum-free Vero cells) — Powder and diluent for suspension for injection Subcutaneous injection
  Arms: vYF
Biological: Yellow fever vaccine — Powder and diluent for suspension for injection Subcutaneous injection
  Other Names: YF-VAX
  Arms: YF-VAX

SUMMARY:
The primary objective of the study is to demonstrate the non-inferiority of the antibody response in terms of seroconversion rate 28 days after vaccine administration of one dose of yellow fever vaccine (vYF) compared to the antibody response after one dose of the YF-VAX control vaccine in yellow fever naïve participants.

The secondary objectives of the study are:

* To describe the immune response to yellow fever in both vaccine groups before and after vYF or YF-VAX administration.
* To describe the safety profile of vYF vaccine in comparison to the safety profile of the control YF-VAX.
* To describe the biosafety profile of vYF in comparison to the biosafety profile of the control YF-VAX.

DETAILED DESCRIPTION:
The duration of each participant's participation will be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 60 years on the day of inclusion.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. A participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) before any dose of study intervention on Day 1 and will be repeated on Day 29 to confirm the participant is still not pregnant within the 28 days of vaccine administration.

* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy, or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known history of flavivirus infection.
* Known systemic hypersensitivity to any of the vaccine components, eggs, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
* Known history or laboratory evidence of human immunodeficiency virus infection.
* Known history of hepatitis B or hepatitis C seropositivity
* Personal or family history of thymic pathology (thymoma, thymectomy, or myasthenia).
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion, including malignancy, such as leukemia, or lymphoma.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Administration of any anti-viral within 2 months preceding the vaccination and up to the 6 weeks following the vaccination
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination except for influenza vaccination, which may be received at least 2 weeks before study vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against a flavivirus disease at any time including YF with either the study vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the past 6 months.
* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the first year of the 5-year follow-up in another clinical study investigating a vaccine, drug, medical device, or medical procedure. Enrollment in another study after the first year is permitted (starting the first day of Year 2, and onwards), assuming it does not exclude participation in this study
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Planned travel in a YF endemic country within 6 months of investigational or control vaccine administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 568 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2027-06-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (11):
- United States (11):
  - Emory University Decatur- Site Number : 8400005, Decatur, Georgia
  - Velocity Clinical Research- New Orleans Site Number : 8400008, New Orleans, Louisiana
  - Johns Hopkins Bloomberg School of Public Health (JHSPH)- Site Number : 8400004, Baltimore, Maryland
  - Harvard University Medical School- Site Number : 8400002, Boston, Massachusetts
  - Saint Louis University- Site Number : 8400003, St Louis, Missouri
  - Meridian Clinical Research- Site Number : 8400009, Omaha, Nebraska
  - SUNY Upstate Medical University Global Health Institute Site Number : 8400006, East Syracuse, New York
  - New York University Langone Medical Center Site Number : 8400013, New York, New York
  - Rochester Clinical Research, Inc.- Site Number : 8400010, Rochester, New York
  - Velocity Clinical Research - Providence Site Number : 8400015, East Greenwich, Rhode Island
  - J Lewis Research Inc- Site Number : 8400012, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 sites in the United States of America from 01 July 2021 to 27 May 2022. Interim results are presented up to Year 2 follow-up, data base lock (DBL) date of 29 August 2024.
Pre-assignment Details: A total of 568 participants were randomized in a 2:1 ratio to receive a single subcutaneous (SC) injection of either yellow fever vaccine (vYF) vaccine or YF-VAX. A subset of participants enrolled at some sites provided an additional post-vaccination blood sample on Day 11 to assess the immune response elicited by both vaccines in terms of neutralizing antibody (NAb) titers and biological safety parameters on Days 1 and 11.
Groups:
- vYF 0.5 mL: Participants received 1 dose of vYF vaccine 0.5 milliliter (mL) as a SC injection on Day 1.
- YF-VAX 0.5 mL: Participants received 1 dose of YF-VAX vaccine 0.5 mL as a SC injection on Day 1.
Period: Overall Study
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Started | 382 | 186
Randomized and Vaccinated | 379 | 186
Completed | 294 | 150
Not Completed | 88 | 36
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Deviation | 4 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 16 | 7
Not completed — Ongoing at the time of DBL date | 60 | 25
Not completed — Randomized but did not receive vaccination | 3 | 0

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants with data in the case report form (CRF).
Groups:
- vYF 0.5 mL: Participants received 1 dose of vYF vaccine 0.5 mL as a SC injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL | Total
Number analyzed (Participants) | 382 | 186 | 568
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.87) | 39.3 (11.88) | 39.7 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 116 | 350
  Male | 148 | 70 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 15 | 12 | 27
  Black or African American | 93 | 53 | 146
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 258 | 112 | 370
  Multiple origin | 6 | 2 | 8
  Not Reported | 5 | 1 | 6
  Unknown | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Yellow Fever (YF)-Naive Participants Who Achieved Seroconversion 28 Days Post Dose 1
Description: Seroconversion was defined as a 4-fold increase in Nab titers as compared to the pre-vaccination value. YF-naive participants (or negative) at baseline corresponded to participants with no detectable YF antibody (Ab) titers before vaccination. The YF NAb titers were determined using a validated live virus microneutralization (MN) assay. Percentages are rounded off to the tenth decimal place.
Time Frame: 28 days post dose 1 (Day 29)
Population: The per-protocol analysis set (PPAS) was a subset of the full analysis set (FAS). The FAS included the subset of randomized participants who received at least 1 dose of the study vaccine or control vaccine and had a valid post-vaccination blood sample result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 329 | 156
percentage of participants | 99.7 [98.3 to 100] | 99.4 [96.5 to 100]
Statistical Analysis 1: Comparison: vYF 0.5 mL vs YF-VAX 0.5 mL; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) was >-5%; Difference in percentage of participants = 0.3, 95% CI 2-sided [-1.2 to 3.2] — 95% CI of the difference was calculated from the Wilson score method without continuity correction

2. Secondary Outcome: Percentage of Participants Who Achieved Seroconversion
Description: Seroconversion was defined as a 4-fold increase in Nab titers as compared to the pre-vaccination value: compared to the Day 1 titers at each timepoint up to Month 6; and to the last planned previous timepoint from Year 1 onwards. The YF NAb titers were determined using a validated live virus MN assay. Percentages are rounded off to the tenth decimal place.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: The FAS included subset of randomized participants who received at least 1 dose of study vaccine or control vaccine and had a valid post-vaccination blood sample result. Day 11: a subset of participants enrolled at some sites provided an additional post-vaccination blood sample on Day 11 to assess the immune response elicited by both vaccines in terms of NAb titers. Only participants with data collected at specified timepoints are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 369 | 183
percentage of participants
  Day 11: number analyzed (Participants) | 59 | 31
  Day 11 | 30.5 [19.2 to 43.9] | 58.1 [39.1 to 75.5]
  Day 29 | 97.8 [95.8 to 99.1] | 98.4 [95.3 to 99.7]
  Month 6: number analyzed (Participants) | 337 | 171
  Month 6 | 94.7 [91.7 to 96.8] | 98.8 [95.8 to 99.9]
  Year 1: number analyzed (Participants) | 315 | 163
  Year 1 | 4.4 [2.5 to 7.3] | 4.9 [2.1 to 9.4]
  Year 2: number analyzed (Participants) | 292 | 150
  Year 2 | 1.4 [0.4 to 3.5] | 1.3 [0.2 to 4.7]

3. Secondary Outcome: Percentage of Participants Who Achieved Seroprotection
Description: Seroprotection was defined as NAb titers >=threshold of 10 (1/dilution). The YF NAb titers were determined using a validated live virus MN assay. Percentages are rounded off to the tenth decimal place.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 371 | 183
percentage of participants
  Day 1 | 6.2 [4.0 to 9.2] | 4.4 [1.9 to 8.4]
  Day 11: number analyzed (Participants) | 59 | 31
  Day 11 | 39.0 [26.5 to 52.6] | 61.3 [42.2 to 78.2]
  Day 29: number analyzed (Participants) | 369 | 183
  Day 29 | 99.5 [98.1 to 99.9] | 99.5 [97.0 to 100]
  Month 6: number analyzed (Participants) | 337 | 171
  Month 6 | 98.8 [97.0 to 99.7] | 99.4 [96.8 to 100]
  Year 1: number analyzed (Participants) | 318 | 163
  Year 1 | 97.5 [95.1 to 98.9] | 97.5 [93.8 to 99.3]
  Year 2: number analyzed (Participants) | 295 | 150
  Year 2 | 98.6 [96.6 to 99.6] | 100 [97.6 to 100]

4. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Yellow Fever Virus
Description: GMTs of antibody against YF virus was measured using a validated live virus MN assay.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 371 | 183
titer
  Day 1 | 5.87 [5.43 to 6.35] | 5.56 [5.11 to 6.05]
  Day 11: number analyzed (Participants) | 59 | 31
  Day 11 | 15.2 [9.69 to 23.7] | 42.6 [20.4 to 88.9]
  Day 29: number analyzed (Participants) | 369 | 183
  Day 29 | 2540 [2218 to 2909] | 3004 [2495 to 3616]
  Month 6: number analyzed (Participants) | 337 | 171
  Month 6 | 544 [467 to 633] | 702 [572 to 861]
  Year 1: number analyzed (Participants) | 318 | 163
  Year 1 | 405 [342 to 480] | 552 [438 to 696]
  Year 2: number analyzed (Participants) | 295 | 150
  Year 2 | 196 [169 to 226] | 245 [200 to 301]

5. Secondary Outcome: Geometric Mean Titers Ratio (GMTRs) of Antibodies Against Yellow Fever Virus
Description: GMTs of antibody against YF virus was measured using a validated live virus MN assay. Ratio was calculated as post-vaccination titer at Days 11, 29 and Month 6 to pre-vaccination titer at Day 1; post-vaccination titer at Year 1 to pre-vaccination titer at Month 6; post-vaccination titer at Year 2 to pre-vaccination titer at Year 1.
Time Frame: Days 1, 11, 29, Month 6, Years 1 and 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 369 | 183
ratio
  Day 11/Day 1: number analyzed (Participants) | 59 | 31
  Day 11/Day 1 | 2.16 [1.49 to 3.12] | 5.57 [2.96 to 10.5]
  Day 29/Day 1 | 227 [194 to 264] | 280 [227 to 344]
  Month 6/Day 1: number analyzed (Participants) | 337 | 171
  Month 6/Day 1 | 49.6 [42.3 to 58.1] | 66.3 [53.7 to 81.8]
  Year 1/Month 6: number analyzed (Participants) | 315 | 163
  Year 1/Month 6 | 0.742 [0.661 to 0.832] | 0.777 [0.658 to 0.916]
  Year 2/Year 1: number analyzed (Participants) | 292 | 150
  Year 2/Year 1 | 0.473 [0.426 to 0.524] | 0.426 [0.367 to 0.495]

6. Secondary Outcome: Number of Participants With Unsolicited Systemic Adverse Events (AEs)
Description: An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, ie, pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to 30 minutes post vaccination on Day 1
Population: The safety analysis set (SafAS) included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 379 | 186
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. An injection site reaction was an AR at and around the injection site of the study vaccine.
Time Frame: Up to 7 days post vaccination (Day 8)
Population: The SafAS included all participants who received at least 1 dose of the study vaccines. Only participants with data collected are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 367 | 185
Participants | 115 | 64

8. Secondary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. Solicited systemic reactions were systemic AEs observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF.
Time Frame: Up to 14 days post vaccination (Day 15)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 367 | 185
Participants | 178 | 102

9. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: as for outcome 6
Time Frame: Up to 28 days post vaccination (Day 29)
Population: The SafAS included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 379 | 186
Participants | 99 | 40

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) up to 6 Months Post-Vaccination
Description: An SAE was any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor could be appropriate. AESIs included serious hypersensitivity/allergic reactions, organ failure/serious viscerotropic events, serious neurologic events.
Time Frame: From the first dose of study vaccine administration (Day 1) up to 6 months post vaccination, approximately up to Day 181
Population: The SafAS included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 379 | 186
Participants
  SAEs | 6 | 2
  AESIs | 0 | 0

11. Secondary Outcome: Number of Participants With Serious Adverse Events and Deaths up to Day 1155
Description: An SAE was any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: From the first dose of study vaccine administration (Day 1) up to DBL date of 29 August 2024, approximately up to Day 1155
Population: The SafAS included all participants who received at least 1 dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 379 | 186
Participants
  SAEs | 6 | 5
  Deaths | 2 | 1

12. Secondary Outcome: Number of Participants With Serious Adverse Events and Deaths Up to Year 5
Description: as for outcome 11
Time Frame: From the first dose of study vaccine administration (Day 1) up to end of study, approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-06

13. Secondary Outcome: Number of Participants With Out-of-Range Biochemistry Parameters
Description: Blood samples were collected at specified timepoints for assessment of biochemistry parameters: alanine aminotransferase (ALT), aspartate transaminase (AST), creatine phosphokinase (CPK), alkaline phosphatase (ALP), bilirubin (accompanied by any increase in liver function test (LFT) and normal LFT), creatinine and C-reactive protein (CRP). The intensity grading scale for laboratory abnormalities was pre-specified in the protocol. Number of participants with out-of-range biochemistry parameters are presented.
Time Frame: Days 1 and 11
Population: Analysis was performed on a subset of participants enrolled at some sites who provided an additional post-vaccination blood sample to assess the biological safety parameters on Days 1 and 11. Only participants with data collected on Days 1 and 11 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 59 | 31
Participants
  Day 1: ALT: number analyzed (Participants) | 55 | 29
  Day 1: ALT | 4 | 0
  Day 11: ALT: number analyzed (Participants) | 58 | 29
  Day 11: ALT | 6 | 1
  Day 1: AST: number analyzed (Participants) | 55 | 29
  Day 1: AST | 3 | 0
  Day 11: AST: number analyzed (Participants) | 59 | 29
  Day 11: AST | 5 | 2
  Day 1: CPK: number analyzed (Participants) | 54 | 28
  Day 1: CPK | 9 | 6
  Day 11: CPK: number analyzed (Participants) | 58 | 31
  Day 11: CPK | 7 | 6
  Day 1: ALP: number analyzed (Participants) | 55 | 29
  Day 1: ALP | 3 | 0
  Day 11: ALP: number analyzed (Participants) | 59 | 30
  Day 11: ALP | 2 | 0
  Day 1: Bilirubin (Any increase in LFT): number analyzed (Participants) | 53 | 28
  Day 1: Bilirubin (Any increase in LFT) | 0 | 0
  Day 11: Bilirubin (Any increase in LFT): number analyzed (Participants) | 59 | 29
  Day 11: Bilirubin (Any increase in LFT) | 0 | 0
  Day 1: Bilirubin (Normal LFT): number analyzed (Participants) | 53 | 28
  Day 1: Bilirubin (Normal LFT) | 1 | 1
  Day 11: Bilirubin (Normal LFT): number analyzed (Participants) | 59 | 29
  Day 11: Bilirubin (Normal LFT) | 1 | 1
  Day 1: Creatinine: number analyzed (Participants) | 55 | 29
  Day 1: Creatinine | 4 | 2
  Day 11: Creatinine | 8 | 2
  Day 1: CRP: number analyzed (Participants) | 48 | 24
  Day 1: CRP | 4 | 4
  Day 11: CRP: number analyzed (Participants) | 52 | 27
  Day 11: CRP | 5 | 4

14. Secondary Outcome: Number of Participants With Out-of-Range Hematology Parameters
Description: Blood samples were collected at specified timepoints for assessment of hematology parameters: red blood cell count (RBC), hematocrit, mean corpuscular volume (MCV), monocytes, basophils, hemoglobin (Hb), white blood cell count (WBC) (increase and decrease), neutrophils and lymphocytes (decrease), eosinophils, platelets (decrease). The intensity grading scale for laboratory abnormalities was pre-specified in the protocol. Number of participants with out-of-range hematology parameters are presented.
Time Frame: Days 1 and 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
Number analyzed (Participants) | 59 | 31
Participants
  Day 1: RBC: number analyzed (Participants) | 55 | 29
  Day 1: RBC | 7 | 4
  Day 11: RBC: number analyzed (Participants) | 59 | 30
  Day 11: RBC | 11 | 5
  Day 1: Hematocrit: number analyzed (Participants) | 55 | 29
  Day 1: Hematocrit | 12 | 6
  Day 11: Hematocrit | 10 | 5
  Day 1: MCV: number analyzed (Participants) | 55 | 29
  Day 1: MCV | 7 | 3
  Day 11: MCV: number analyzed (Participants) | 59 | 30
  Day 11: MCV | 5 | 2
  Day 1: Monocytes: number analyzed (Participants) | 51 | 28
  Day 1: Monocytes | 6 | 1
  Day 11: Monocytes: number analyzed (Participants) | 51 | 29
  Day 11: Monocytes | 6 | 4
  Day 1: Basophils: number analyzed (Participants) | 47 | 27
  Day 1: Basophils | 0 | 0
  Day 11: Basophils: number analyzed (Participants) | 47 | 27
  Day 11: Basophils | 0 | 0
  Day 1: Hb: number analyzed (Participants) | 55 | 29
  Day 1: Hb | 12 | 7
  Day 11: Hb | 10 | 6
  Day 1: WBC increase: number analyzed (Participants) | 55 | 29
  Day 1: WBC increase | 2 | 1
  Day 11: WBC increase: number analyzed (Participants) | 59 | 30
  Day 11: WBC increase | 13 | 0
  Day 1: WBC decrease: number analyzed (Participants) | 55 | 29
  Day 1: WBC decrease | 2 | 1
  Day 11: WBC decrease: number analyzed (Participants) | 59 | 30
  Day 11: WBC decrease | 13 | 0
  Day 1: Neutrophils decrease: number analyzed (Participants) | 51 | 29
  Day 1: Neutrophils decrease | 2 | 1
  Day 11: Neutrophils decrease: number analyzed (Participants) | 51 | 29
  Day 11: Neutrophils decrease | 8 | 3
  Day 1: Lymphocytes decrease: number analyzed (Participants) | 51 | 29
  Day 1: Lymphocytes decrease | 0 | 0
  Day 11: Lymphocytes decrease: number analyzed (Participants) | 51 | 29
  Day 11: Lymphocytes decrease | 2 | 1
  Day 1: Eosinophils: number analyzed (Participants) | 51 | 29
  Day 1: Eosinophils | 1 | 2
  Day 11: Eosinophils: number analyzed (Participants) | 51 | 29
  Day 11: Eosinophils | 1 | 2
  Day 1: Platelets decrease: number analyzed (Participants) | 55 | 29
  Day 1: Platelets decrease | 4 | 1
  Day 11: Platelets decrease | 5 | 0

ADVERSE EVENTS:
Time Frame: AEs, SAEs and all-cause mortality (deaths) were collected from the first dose of study vaccine administration (Day 1) up to DBL date of 29 August 2024, approximately up to Day 1155
Description: Analysis was performed on the SafAS. Interim results are presented up to Year 2 follow-up, DBL date of 29 August 2024.
Arm/Group | vYF 0.5 mL | YF-VAX 0.5 mL
All-Cause Mortality (participants affected / at risk) | 2/379 | 1/186
Serious Adverse Events (participants affected / at risk) | 6/379 | 5/186
Other Adverse Events (participants affected / at risk) | 206/379 | 113/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vYF 0.5 mL (N=379) | YF-VAX 0.5 mL (N=186)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vYF 0.5 mL (N=379) | YF-VAX 0.5 mL (N=186)
Injection Site Erythema (General disorders) | 27 (27) | 8 (8)
Injection Site Pain (General disorders) | 105 (105) | 58 (58)
Malaise (General disorders) | 110 (110) | 63 (63)
Myalgia (Musculoskeletal and connective tissue disorders) | 114 (114) | 59 (59)
Headache (Nervous system disorders) | 134 (134) | 70 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04942210/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT04942210/SAP_001.pdf